CLINICAL TRIAL: NCT05192655
Title: Künstliche Intelligenz (KI) in Der Funktionellen Bildgebung Zur Individualisierten Behandlung Von Kopf-Hals-Plattenepithelkarzinom-Patienten Artificial Intelligence in Functional Imaging for Individualized Treatment of Head and Neck Squamous Cell Carcinoma Patients
Brief Title: Artificial Intelligence in Functional Imaging for Individualized Treatment of Head and Neck Squamous Cell Carcinoma Patients
Acronym: KIVAL-KHT
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Helmholtz-Zentrum Dresden-Rossendorf (Unknown); Max-Delbrück-Centrum Berlin (Unknown)
Responsible Party: Principal Investigator, Julian Weingärtner, Resident at the Department of Radiooncology and Radiotherapy, Charité; BIH Charité Junior Digital Clinician Scientist, Charite University, Berlin, Germany
Other Study IDs: KIVAL-KHT
Record Dates: First submitted 2021-12-14; First posted 2022-01-14 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Analysis of genome sequences for risk stratification planned in further studies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HNSCC-patients treated with primary radio(chemo)therapy (R(C)T): Patients, older than 18 years, with diagnosed HNSCC, attending the Department of Radiooncology and Radiotherapy at Charité for a treatment with curative intension (R(C)T) . All patients received as pretherapeutic diagnostic method a 18F-Fluorodesoxyglucose (FDG) positron emission tomography (PET) imaging.
  Interventions: Other: Observation
- HNSCC-patients treated with primary surgery: Patients, older than 18 years, with diagnosed HNSCC, attending the Department of Oral and Maxillofacial Surgery or ENT Department at Charité for a treatment with curative intension ( primary surgery +/- combined with adjuvant (R(C)T)). All patients received as pretherapeutic diagnostic method a 18F-Fluorodesoxyglucose (FDG) positron emission tomography (PET) imaging.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation Study

SUMMARY:
The two curative treatment modalities for patients with HNSCC - primary chemoradiation (CRT) or primary surgery (often combined with postoperative (C)RT) - are both associated with serious side effects for which reason further stratification, optimization and personalization of treatment is urgently needed. As novel quantitative image analyses are a promising tool for further risk stratification, the investigators training a three-dimensional Convolutional Neural Network on 18F-Fluorodesoxyglucose (FDG) positron emission tomography (PET) imaging and clinical / histopathological data of a multicentric, retrospective cohort of 1200 patients treated with primary CRT and 800 patients treated with primary surgery at Charité and cooperation institutes in order to predict individual treatment-specific outcomes and identify patients with excellent outcome after primary CRT or primary surgery or unfavorable outcome for both. The trained algorithm of the artificial intelligence will be validated in a prospective trial to see if predicted loco-regional control and recommended treatment strategies are reliable. In total 250 curative HNSCC patients, treated with CRT or primary surgery, will be enrolled on this prospective validation trial with observational character, while biomarker, clinical and FDG-PET data are collected from these patients and follow-up visits will be concluded.

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 18 years with diagnosed HNSCC, attending the Department of Radiooncology and Radiotherapy or the Department of Oral and Maxillofacial Surgery at Charité for a treatment with curative intension ( R(C)T or primary surgery / combined).
* All patients received as pretherapeutic diagnostic method a 18F-Fluorodesoxyglucose (FDG) positron emission tomography (PET) imaging

Exclusion Criteria:

* Patients with HNSCC who cannot be treated in a curative approach
* Patients with HNSCC treated in a curative approach but unable to receive FDG PET imaging before start of treatment
* Data from patients who have withdrawn their study consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years with diagnosed HNSCC, attending the Department of Radiooncology and Radiotherapy or the Department of Oral and Maxillofacial Surgery at Charité for a treatment with curative intension ( primary R(C)T or primary surgery / combined).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Locoregional Control | 2 years
  Freedom from local progression within the first two years after treatment. Failure of locoregional control is defined as relapse of tumor confirmed by biopsy or if biopsy is inadequate or not feasible, consisting clear image morphology (MRI / CT / PET) during routine follow-up check-ups

SECONDARY OUTCOMES:
Life Quality | 2 years
  Collection of questionares regarding life quality before treatment and during routine follow-up check-ups after treatment regarding to the European Quality of Life Instrument (EURO-QOL)
Metastases-free survival | 2 years
  Freedom of Metastasis within the first two years after treatment during routine follow-up check-ups; Metastasis must be confirmed by biopsy or clear image morphology if a biopsy is not feasible (MRI / CT / PET)
Toxicity of Treatment | 2 years
  Collection of questionares regarding toxicity according to Common Toxicity Criteria (CTC) during routine follow-up check-ups
Progression-free Survival | 2 years
  alternative for Overall survival; event in PFS defined as disease progression or death

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiooncology and Radiotherapy, Charité - Universitätsmedizin Berlin, Campus Virchow Klinikum, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
In order to enable a replication by independent researchers, the AI technology and algorithm will be made publicly accessible. Patients of the prospective imaging trial have the option to consent to the pseudonymized publication of their imaging data, this enables upload of the dataset to public image repositories. In this way the reproduction and thus verification of the results of the prospective part will be possible. Imaging protocols, analyzed scans, details about the extracted features and of the modelling and segmentation methodology will be disclosed.